CLINICAL TRIAL: NCT04315909
Title: A Randomized, Double-Blind, Parallel-group, Clinical Trial to Evaluate the Effect of Platelet-Rich Plasma-Fibrin Glue in Combination With Vitamin E and C for Treatment of Non-healing Diabetic Foot Ulcers
Brief Title: The Effect of Platelet-Rich Plasma-Fibrin Glue in Combination With Vitamin E and C for Treatment of Non-healing Diabetic Foot Ulcers
Status: Unknown | Phase: Phase 2 / Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Mashhad University of Medical Sciences (Other)
Responsible Party: Principal Investigator, Daryoush Hamidi Alamdari, Associate professor, Mashhad University of Medical Sciences
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: IR.MUMS.REC.1398.125
Record Dates: First submitted 2020-03-17; First posted 2020-03-20 (Actual); Last update posted 2020-03-20 (Actual); Status verified 2020-03

CONDITIONS: Diabetic Foot Ulcers; Diabetic Wound
Keywords: Platelet-Rich Plasma-Fibrin Glue; DFU; Vitamin E; Vitamin C; non-healing Diabetic Foot Ulcers
MeSH Terms: conditions — Diabetic Foot | interventions — Vitamin E

STUDY DESIGN:
Who Masked: Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention group (Experimental): Patients with non-healing Diabetic Foot Ulcers treated with PRP-Fibrin-Glue plus vitamin supplements (E (200 IU/ 2day) and C (250 mg/ 2day) ) for 8 weeks.
  Interventions: Drug: PRP-Fibrin Glue; Dietary Supplement: Vitamin E and C
- Control group (Experimental): Patients with non-healing Diabetic Foot Ulcers treated with PRP-Fibrin-Glue plus placebo for 8 weeks.
  Interventions: Drug: PRP-Fibrin Glue; Other: Placebo

INTERVENTIONS:
Drug: PRP-Fibrin Glue — Platelet-Rich Plasma-Fibrin Glue
  Other Names: Platelet-Rich Plasma-Fibrin Glue
Dietary Supplement: Vitamin E and C — Vitamin E and vitamin C
  Arms: Intervention group
Other: Placebo — Placebo
  Arms: Control group

SUMMARY:
The aim of this study is to evaluates the chance of non-healing Diabetic Foot Ulcers repair by reducing oxidative stress caused by diabetes by taking vitamin E and C supplements along with the use of Platelet-Rich Plasma-Fibrin Glue as an effective treatment for wound healing.

ELIGIBILITY:
Inclusion Criteria:

1. DFU is classified as Wagner 1 -2 on the Wagner classification system.
2. Persons with type 1 or type 2 diabetes with a non-healing ulcer of at least 4 weeks duration.
3. If more than one non-healing wound is present, the largest of the wounds that is classified as a Wagner 1- 2.
4. The index ulcer had to be clinically non-infected.
5. Ankle Brachial Index (ABI) greater than or equal to 0.7.
6. HemoglobinA1C (HbA1c) < 12
7. Index foot ulcer located on the plantar, medial, or lateral aspect of the foot (including all toe surfaces).
8. Wound area (length x width) measurement between 2 cm2 and 20 cm2.
9. Non-use of drugs that may interfere with wound healing, such as corticosteroids, immunosuppressive agents, and cytotoxic agents.
10. No smoking, alcohol or drug addiction.
11. Approved, informed, signed consent.

Exclusion Criteria:

1. Previous consumption of vitamin E and C supplements.
2. Index ulcer has exposed tendons, ligaments, muscle, or bone.
3. Confirmed presence of osteomyelitis, or if osteomyelitis is suspected.
4. Patients with renal deficiency, hepatic failure, has known immune insufficiency and cancer.
5. Subject is pregnant or plans to become pregnant during the duration of the trial.
6. Patient's blood vessels are non-compressible for ABI testing.
7. Patient is known to have a psychological, developmental, physical, emotional disorders.
8. Received systemic corticosteroids or immunosuppressive agents.

Ages: 35 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Estimated)
Dates: Start 2019-08-28 (Actual); Primary Completion 2020-06-23 (Estimated); Study Completion 2020-06-23 (Estimated)

PRIMARY OUTCOMES:
Healing rate of the ulcer | 2 months
  Examination by a vascular surgery physician and documentation
Wound Size | 2 months
  Wound size will be measured with ruler for length, width as well as with digital imaging. Wound size will be assessed in digital images taken of the wound.

SECONDARY OUTCOMES:
Serum ESR at baseline and after the intervention | 2 months
  Erythrocyte Sedimentation Rate
Serum hs-CRP at baseline and after the intervention | 2 months
  high-sensitivity C-Reactive Protein
FBS at baseline and after the intervention | 2 months
  Fasting blood sugar
HbA1c at baseline and after the intervention | 2 months
  Glycated hemoglobin
Lipid Profile at baseline and after the intervention | 2 months
  Serum Triglyceride, Cholesterol, HDL, LDL, VLDL
Serum Urea at baseline and after the intervention | 2 months
  In a quantitative laboratory method
Serum Creatinine at baseline and after the intervention | 2 months
  In a quantitative laboratory method
Serum total bilirubin at baseline and after the intervention | 2 months
  In a quantitative laboratory method
Serum Uric acid at baseline and after the intervention | 2 months
  In a quantitative laboratory method
Serum Homocysteine at baseline and after the intervention | 2 months
  In a quantitative laboratory method
Pro-Oxidant Antioxidant Balance at baseline and after the intervention | 2 months
  The PAB assay is a test to determine the oxidants and antioxidants simultaneously in one single test.

CONTACTS AND LOCATIONS:
Overall Officials: Daryoush Hamidi Alamdari, Ph.D, Principal Investigator — Mashhad University of Medical Sciences, Mashhad, Iran
Locations (1):
- Alavi Hospital, Mashhad, Razavi Khorasan Province, Iran

IPD SHARING:
Plan to Share IPD: Yes
All data related to the project after unidentifiable of people will be shared.
Supporting Information: Study Protocol, ICF
Time Frame: Access to data are allowed 6 months after the publication of results.
Access Criteria: The investigator's data will be available for university staffs and academic institutions.

REFERENCES:
- [Derived] Yarahmadi A, Saeed Modaghegh MH, Mostafavi-Pour Z, Azarpira N, Mousavian A, Bonakdaran S, Jarahi L, Samadi A, Peimani M, Hamidi Alamdari D. The effect of platelet-rich plasma-fibrin glue dressing in combination with oral vitamin E and C for treatment of non-healing diabetic foot ulcers: a randomized, double-blind, parallel-group, clinical trial. Expert Opin Biol Ther. 2021 May;21(5):687-696. doi: 10.1080/14712598.2021.1897100. Epub 2021 Apr 13. PMID 33646060